CLINICAL TRIAL: NCT02933489
Title: Comparison of Abbreviated Breast MRI and Digital Breast Tomosynthesis in Breast Cancer Screening in Women With Dense Breasts
Brief Title: Abbreviated Breast MRI and Digital Tomosynthesis Mammography in Screening Women With Dense Breasts
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: EA1141; NCI-2016-00252 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s16-01825 (Other: Other); EA1141 (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EA1141 (Other: DCP); EA1141 (Other: CTEP); UG1CA189828 (NIH)
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Asymptomatic
MeSH Terms: interventions — Dynamic Contrast Enhanced Magnetic Resonance Imaging; Mammography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm A (DBT, AB-MR) (Experimental): Participants undergo DBT followed by AB-MR for under 10 minutes on the same day or within 24 hours at baseline and then after 1 year.
  Interventions: Diagnostic Test: Contrast-enhanced Magnetic Resonance Imaging; Diagnostic Test: Digital Tomosynthesis Mammography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (AB-MR, DBT) (Experimental): Participants undergo AB-MR for under 10 minutes followed by DBT on the same day or within 24 hours at baseline and then after 1year.
  Interventions: Diagnostic Test: Contrast-enhanced Magnetic Resonance Imaging; Diagnostic Test: Digital Tomosynthesis Mammography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced Magnetic Resonance Imaging — Undergo AB-MR
  Other Names: CONTRAST ENHANCED MRI; Contrast-enhanced MRI
Diagnostic Test: Digital Tomosynthesis Mammography — Undergo DBT
  Other Names: DBT; Digital Breast Tomosynthesis; Digital Tomosynthesis of the Breast
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well abbreviated breast magnetic resonance imaging (MRI) and digital tomosynthesis mammography work in detecting cancer in women with dense breasts. Abbreviated breast MRI is a low cost procedure in which radio waves and a powerful magnet linked to a computer and used to create detailed pictures of the breast in less than 10 minutes. These pictures can show the difference between normal and diseased tissue. Digital tomosynthesis mammography is a procedure that uses multiple x-rays pictures of each breast to produce a 3-dimensional rendering of the entire breast. Combined screening with abbreviated breast MRI and digital tomosynthesis mammography may be a better method to screen women with dense breasts.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the rates of detection of invasive cancers between the initial abbreviated breast (AB)-magnetic resonance (MR) and digital tomosynthesis mammography (DBT).

SECONDARY OBJECTIVES:

I. To compare the positive predictive value (PPV) of biopsies, call back rates, and short-term follow up rates after AB-MR and DBT on both the initial and 1 year follow up studies.

II. To estimate and compare the sensitivity and specificity of AB-MR and DBT, using the 1 year follow up to define a reference standard.

III. To compare patient-reported short-term quality of life related to diagnostic testing with AB-MR and DBT using the Testing Morbidities Index.

IV. To compare willingness to return for testing with AB-MRI versus (vs) DBT within the recommended screening interval and explore factors associated with willingness to return for screening.

V. To compare the tumor biologies of invasive cancers and ductal carcinoma in situ (DCIS) detected on AB-MR and DBT.

VI. To estimate the incident cancer rate during 3 years following the year-1 AB-MR/DBT when patients return to standard screening.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A (DBT, AB-MR): Participants undergo DBT followed by AB-MR for under 10 minutes on the same day or within 24 hours at baseline and then after 1 year.

ARM B (AB-MR, DBT): Participants undergo AB-MR for under 10 minutes followed by DBT on the same day or within 24 hours at baseline and then after 1 year.

After completion of study, patients are followed up at every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patents must be scheduled for routine screening DBT
* Women must not be pregnant or breast-feeding; all females of childbearing potential who are uncertain if they could be pregnant or may be pregnant or as per local site standard of practice in women undergoing DBT and MRI must have a blood test or urine study within 2 weeks prior to randomization to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the following year until the year 1 AB-MR and DBT studies are performed
* Patient?s breast density must be known; patients must have mammographically dense breasts, American College of Radiology [ACR] Breast Imaging [BI]- Reporting and Data System Atlas (RADS) lexicon categories c or d (heterogeneous or extreme fibroglandular tissue) on their most-recent prior screening
* Patient must be asymptomatic for breast disease and undergoing routine screening
* Patient must have no known breast cancer (DCIS or invasive cancer), not currently undergoing treatment for breast cancer, or planning surgery for a high risk lesion (atypical ductal breast hyperplasia [ADH], atypical lobular breast hyperplasia [ALH], lobular breast carcinoma in situ [LCIS], papilloma, radial scar)
* Patient must not be taking chemoprevention for breast cancer
* Patient must not have undergone breast ultrasound within 12 months prior to randomization
* Patient must not have previously had a breast MRI
* Patient must not have previously had molecular breast imaging (MBI, multiplexed ion beam imaging [MIBI])
* Patient must agree to not undergo screening ultrasound (of breast) for the duration of the 1 year study period
* Patient must not be suspected of being at high-risk for breast cancer, as defined by the American Cancer Society (ACS) breast MR screening recommendations (lifetime risk of >= 20-25%)
* Patient must be able to undergo breast MRI with contrast enhancement; patients unable to undergo breast MRI with contrast enhancement for any reason are ineligible

  * No history of untreatable claustrophobia
  * No presence of non MR compatible metallic objects or metallic objects that, in the opinion of the radiologist, would make MRI a contraindication
  * No history of sickle cell disease
  * No contraindication to intravenous contrast administration
  * No known allergy-like reaction to gadolinium or moderate or severe allergic reactions to one or more allergens as defined by the American College of Radiology (ACR); patient may be eligible if willing to undergo pre-treatment as defined by the institution's policy and/or ACR guidance
  * No known or suspected renal impairment; requirements for glomerular filtration rate (GFR) prior to MRI as determined by local site standard practice
  * Weight less than or equal to the MRI table limit
  * No women who have had prior contrast enhanced mammography (contrast enhanced spectral mammography [CESM] or contrast enhanced digital mammography [CEDM])
  * No women who have breast prosthetic implants (silicone or saline) Exclusion Criteria

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1516 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Comstock, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (68):
- United States (67):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Huntington Memorial Hospital, Pasadena, California
  - The Women's Imaging Center, Denver, Colorado
  - Radiology Imaging Associates, Englewood, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Diagnostic Center for Women LLC, Miami, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Clinical Radiologists SC, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Aultman Health Foundation, Canton, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
- Rwth Klinikum Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Safe harbor de-identified data corresponding to publications will be shared upon request
Supporting Information: Study Protocol, SAP
Time Frame: With publication
Access Criteria: All requests will require a statistical plan and justification. Approved requests will require a DUA.
URL: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7276668/bin/NIHMS1578579-supplement-Supplement_I.docx

REFERENCES:
- [Result] Comstock CE, Gatsonis C, Newstead GM, Snyder BS, Gareen IF, Bergin JT, Rahbar H, Sung JS, Jacobs C, Harvey JA, Nicholson MH, Ward RC, Holt J, Prather A, Miller KD, Schnall MD, Kuhl CK. Comparison of Abbreviated Breast MRI vs Digital Breast Tomosynthesis for Breast Cancer Detection Among Women With Dense Breasts Undergoing Screening. JAMA. 2020 Feb 25;323(8):746-756. doi: 10.1001/jama.2020.0572. PMID 32096852
- See also: Primary Manuscript — https://pubmed.ncbi.nlm.nih.gov/32096852/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women with dense breasts scheduled for routine screening with DBT were enrolled to receive DBT and AB-MR, with scan order determined by randomization. The first subject was accrued on December 27, 2016, and accrual ended on November 10, 2017. A total of 48 institutions participated.
Groups:
- Arm A (DBT, AB-MR): Participants undergo DBT followed by AB-MR, for under 10 minutes, on the same day or within 24 hours at baseline and then after 1 year.
  AB-MR: Contrast-enhanced Abbreviated Magnetic Resonance Imaging (MRI) DBT: Digital Tomosynthesis Mammography
- Arm B (AB-MR, DBT): Participants undergo AB-MR, for under 10 minutes, followed by DBT on the same day or within 24 hours at baseline and then after 1 year.
  AB-MR: Contrast-enhanced Abbreviated Magnetic Resonance Imaging (MRI) DBT: Digital Tomosynthesis Mammography
Period: Overall Study
Arm/Group | Arm A (DBT, AB-MR) | Arm B (AB-MR, DBT)
Started | 757 | 759
DBTperformed | 726 | 737
AB MR Performed | 713 | 733
DCIS Detected | 5 | 6
PAM50 NanoString | 0 | 0
Completed | 713 | 731
Not Completed | 44 | 28
Not completed — Ineligible | 3 | 3
Not completed — Withdrawal by Subject | 27 | 18
Not completed — Unable to complete exams (other) | 14 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (DBT, AB-MR) | Arm B (AB-MR, DBT) | Total
Number analyzed (Participants) | 757 | 759 | 1516
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (8.7) | 54.9 (8.4) | 54.9 (8.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 757 | 759 | 1516
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 31 | 42
  Not Hispanic or Latino | 704 | 678 | 1382
  Unknown or Not Reported | 42 | 50 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 38 | 22 | 60
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 29 | 41 | 70
  White | 648 | 639 | 1287
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 41 | 53 | 94
Menopausal Status [Count of Participants; unit: Participants]
  Pre-menopausal | 236 | 206 | 442
  Peri-menopausal | 49 | 45 | 94
  Naturally post-menopausal | 316 | 355 | 671
  Surgically post-menopausal | 114 | 129 | 243
  Unknown (data not available) | 42 | 24 | 66
Breast density (baseline DBT) [Count of Participants; unit: Participants]
  Almost entirely fat | 1 | 1 | 2
  Scattered fibroglandular densities | 50 | 66 | 116
  Heterogeneously dense | 564 | 564 | 1128
  Extremely dense | 113 | 109 | 222
  Scan not performed | 29 | 19 | 48
Prior personal history of breast cancer [Count of Participants; unit: Participants]
  No | 724 | 728 | 1452
  Yes | 3 | 6 | 9
  Unknown | 30 | 25 | 55

OUTCOME MEASURES:

1. Primary Outcome: Screen-detected Invasive Cancer Verified by Pathology
Description: For each modality, the detection rate of invasive cancers is defined as the proportion of participants who had an invasive cancer detected by the modality at baseline and verified by pathology versus the total number of participants. In the out come measures table below, these proportions will be automatically calculated, multiplied by 100, and be presented as percentages (%).
Time Frame: Up to 1 year
Population: Subjects with both DBT and AB-MR
Measure: Count of Participants; unit: Participants
Groups:
- Digital Breast Tomosynthesis (DBT): Detection of Cancer based on results of Digital Breast Tomosynthesis (DBT) performed within 30 days following registration.
  DBT and abbreviated -MR were performed on the same day and interpreted by two different radiologists, each blinded to the other modality. However, DBT and AB-MR were allowed to be performed within 24 hours of each other, as long as the radiologists remained blinded to the results of the other modality
- Abbreviated Breast MR (AB-MR): Detection of Cancer based on results of abbreviated breast MR (AB-MR) performed within 30 days following registration.
  DBT and AB-MR were performed on the same day and interpreted by two different radiologists, each blinded to the other modality. However, DBT and AB-MR were allowed to be performed within 24 hours of each other, as long as the radiologists remained blinded to the results of the other modality
Arm/Group | Digital Breast Tomosynthesis (DBT) | Abbreviated Breast MR (AB-MR)
Number analyzed (Participants) | 1444 | 1444
Participants
  No Invasive Cancer Detected | 1437 | 1427
  Invasive Cancer Detected | 7 | 17
Statistical Analysis 1: Comparison: Digital Breast Tomosynthesis (DBT) vs Abbreviated Breast MR (AB-MR); The proportion of participants who had an invasive cancer, verified by pathology, detected by each modality (the invasive cancer detection rates) will be made using exact McNemar's test; Test type: Equivalence — H0: DBT = AB-MR; p = 0.002, McNemar; Wald interval with Bonett-Price Laplace = 0.007, 95% CI 2-sided [0.0022 to 0.0116] — Wald interval with Bonett-Price Laplace, described in : Fagerland MW, Lydersen S, Laake P. Recommended tests and confidence intervals for paired binomial proportions. Statist. Med. 2014; 33:2850-75

2. Secondary Outcome: Positive Predictive Value (PPV) of Biopsies
Description: Test Positive (T+): Biopsy recommended by imaging, defined as patients with at least one lesion rated BI-RADS 4 or 5 on image interpretation. Reference Standard Positive (RS+): Pathologically confirmed DCIS or invasive disease resultant from a positive test.
  The 95% confidence interval for PPV of biopsy for each modality were derived from the GEE model using the appropriate estimable contrasts with robust standard errors
Time Frame: Baseline to up to 1 year
Population: Positive predictive value is calculated on patients with at least one lesion rated BI-RADS 4 or 5 on image interpretation (I.e., Biopsy recommended) and is the percentage of biopsy recommended by imaging test versus patients with cancer P(D+|T+)
Measure: Number (95% Confidence Interval); unit: percentage of Biopsy Recommended
Units Other Than Participants: Cases recommended for biopsy by imaging
Groups:
- Biopsy Recommended by Digital Breast Tomography: Patients with at least one lesion rated BI-RADS 4 or 5 on image interpretation.
- Biopsy Recommended by AB-MR: Patients with at least one lesion rated BI-RADS 4 or 5 on Abbreviated MR interpretation.
Arm/Group | Biopsy Recommended by Digital Breast Tomography | Biopsy Recommended by AB-MR
Number analyzed (Participants) | 1444 | 1444
Number analyzed (Cases recommended for biopsy by imaging) | 29 | 107
percentage of Biopsy Recommended | 31.0 [17.0 to 49.7] | 19.6 [13.2 to 28.2]
Statistical Analysis 1: Comparison: Biopsy Recommended by Digital Breast Tomography vs Biopsy Recommended by AB-MR; Positive Predictive Value (PPV); Test type: Equivalence — PPV DBT = PPV AB-MR; p = 0.15, Leisenring — Generalized estimating equation (GEE) regression with the p-value from the resulting score test. 5 secondary comparisons were planned: alpha level of 0.05/5 = 0.01 for p-value significance; Leisenring W, Alonzo T, Pepe MS. Comparisons of predictive values of binary medical diagnostic tests for paired designs. Biometrics. 2000;56:345-351

3. Secondary Outcome: Call Back/Additional Imaging/Short-term Follow Rates for DBT and AB-MR
Description: For DBT:
  DBT: Call back is defined as having additional views or targeted ultrasound to evaluate DBT findings DBT: short term follow up (STFU) is defined as having at least one lesion rated BI-RADS 3 on DBT DBT: Additional imaging recommendation is defined as having either call back or STFU
  For AB-MR:
  Ab-MR: Call back does not apply to AB-MR and will not be evaluated Ab-MR: Short Term Follow-up (STFU) is defined as having at least one lesion rated BI-RADS 3 on AB-MR Ab-MR: Additional imaging recommendation is defined as having a STFU
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- DBT Additional Imaging Recommendation: subjects requiring further assessment by DBT (i.e. either a call back or short term follow up (STFU)) Call back is defined as having additional views or targeted ultrasound to evaluate DBT findings STFU is defined as having at least one lesion rated BI-RADS 3 on DBT Additional imaging recommendation is defined as having either call back or STFU
- AB-MR Additional Imaging Recommendation: subjects requiring further assessment by AB-MR Call back does not apply to AB-MR and will not be evaluated Short Term Follow-up (STFU) is defined as having at least one lesion rated BI-RADS 3 on AB-MR Additional imaging recommendation is defined as having a STFU
Arm/Group | DBT Additional Imaging Recommendation | AB-MR Additional Imaging Recommendation
Number analyzed (Participants) | 1444 | 1444
Participants
  Call back | 146 | NA — For AB-MR, the definition of call back does not apply.
  Short-term follow-up (subject-level) | 18 | 108
  Additional imaging recommendation | 146 | 108
Statistical Analysis 1: Comparison: DBT Additional Imaging Recommendation vs AB-MR Additional Imaging Recommendation; The exact p-value from McNemar's test is reported for for comparing the DBT against the AB-MR short term follow-up rates; Test type: Equivalence — H0: DBT short term follow-up rate = AB-MR short term follow-up rate; p < 0.0001, McNemar — To adjust for multiplicity, using the Bonferroni correction, secondary comparisons are compared against an adjusted alpha level of 0.05/5=0.01 corresponding to the 5 secondary comparisons outlined in the Statistical Analysis Plan (SAP); exact p-value
Statistical Analysis 2: Comparison: DBT Additional Imaging Recommendation vs AB-MR Additional Imaging Recommendation; The exact p-value from McNemar's test is reported for for comparing the DBT against the AB-MR additional imaging rates; Test type: Equivalence — H0: DBT additional imaging rate =AB-MR additional imaging rate; p = 0.02, McNemar — To adjust for multiplicity, using the Bonferroni correction, secondary comparisons are compared against an adjusted alpha level of 0.05/5 = 0.01, corresponding to the 5 secondary comparisons outlined in the SAP; exact p-values

4. Secondary Outcome: Prediction of Breast Cancer (Sensitivity and Specificity)
Description: Reference standard positive (RS+): breast cancer (invasive or DCIS) detected on the year 0 screening or reported at any time from the year 0 to the year 1 screening.
  Reference standard negative (RS-): No breast cancer reported at any time from the year 0 to the year 1 screen.
  Incomplete: No Year 1 imaging, and <11 months of patient follow-up (<330 days) after year 0 screen
  Positive Test (T+) is defined as the imaging modality result is positive (BI-RADS 3-5), and the location of the finding is matches the location of the cancer indicated by the reference standard.
  Negative Test (T-) will be estimated as the fraction of reference standard negative subjects for whom the imaging modality result was negative (BI-RADS 1-2).
  95% confidence intervals for the sensitivity and specificity of each modality calculated using the Wilson method.
Time Frame: Baseline to up to 1 year
Population: of the 1444 women available for analysis 14 were missing reference standard information.
Measure: Number (95% Confidence Interval); unit: percentage of correct classifications
Groups:
- Test A: Digital Breast Tomography: Results of the Digital Breast Tomography (DBT) interpretation
- Test B: Abbreviated MR: Results of the Abbreviated MR interpretation
Arm/Group | Test A: Digital Breast Tomography | Test B: Abbreviated MR
Number analyzed (Participants) | 1430 | 1430
percentage of correct classifications
  Sensitivity (T+|RS+): number analyzed (Participants) | 23 | 23
  Sensitivity (T+|RS+) | 39.1 [22.2 to 59.2] | 95.7 [79.0 to 99.2]
  Specificity (T-|RS-): number analyzed (Participants) | 1407 | 1407
  Specificity (T-|RS-) | 97.4 [96.5 to 98.1] | 86.7 [84.8 to 88.4]
Statistical Analysis 1: Comparison: Test A: Digital Breast Tomography vs Test B: Abbreviated MR; Test type: Equivalence — Sensitivity DBT = Sensitivity AB-MR; p = 0.001, McNemar — The comparison of the sensitivity of AB-MR and DBT uses a two-sided exact McNemar's test to account for the paired design 5 secondary comparisons were planned: alpha level of 0.05/5 = 0.01 for p-value significance
Statistical Analysis 2: Comparison: Test A: Digital Breast Tomography vs Test B: Abbreviated MR; Test type: Equivalence — Specificity DBT = Specificity AB-MR; p < 0.001, McNemar — The comparison of the Specificity of AB-MR and DBT uses a two-sided exact McNemar's test to account for the paired design 5 secondary comparisons were planned: alpha level of 0.05/5 = 0.01 for p-value significance

5. Secondary Outcome: Change in Patient-reported Short-term Quality of Life Related to Diagnostic Testing
Description: Testing Morbidities Index (TMI) scores [0 (worst) to 100 (best) scale] will be computed for abbreviated breast-magnetic resonance (MR) and digital tomosynthesis mammography (DBT) after the baseline screen.
Time Frame: Baseline to up to 1 year
Population: Participants with both DBT and MRI performed and completed PRO surveys
Measure: Mean (95% Confidence Interval); unit: score on 0-100 scale
Groups:
- Abbreviated MRI: Subjects with Abbreviated MRI and completed PRO surveys.
- Digital Breast Tomosynthesis: Subjects with Digital Breast Tomosynthesis and completed PRO surveys.
Arm/Group | Abbreviated MRI | Digital Breast Tomosynthesis
Number analyzed (Participants) | 1321 | 1321
score on 0-100 scale
  TMI component during exam | 90.1 [89.5 to 90.7] | 86.3 [85.6 to 86.9]
  TMI component after exam | 98.4 [98.0 to 98.7] | 99.0 [98.7 to 99.3]

6. Secondary Outcome: Willingness to Return for Testing With Abbreviated Breast-magnetic Resonance (MR) Versus Digital Tomosynthesis Mammography (DBT)
Description: The proportions of participants willing to return for screening with either test, AB-MRI only, DBT only, or not willing to return for either test will be estimated.
Time Frame: Up to 1 year
Population: Subjects with AB-MR, DBT and completed surveys
Measure: Count of Participants; unit: Participants
Groups:
- Abbreviated MRI Willingness to be Screened in the Future: Subjects with Abbreviated MRI and completed PRO surveys and their willingness to be screened in the future
- Digital Breast Tomosynthesis Willingness to be Screened in the Future: Subjects with Digital Breast Tomosynthesis and completed PRO surveys and their willingness to be screened in the future
- Ab-MRI Future Screen if AB-MRI Detects More Cancer Than Mammography or Ultrasound: Subjects with Abbreviated MRI and completed PRO surveys and their willingness to be screened in the future if AB-MRI Detects More Cancer than Mammography or Ultrasound
- DBT Future Screen if DBT Detects More Cancer Than Mammography or Ultrasound: Subjects with DBT and completed PRO surveys and their willingness to be screened in the future if DBTDetects More Cancer than Mammography or Ultrasound
Arm/Group | Abbreviated MRI Willingness to be Screened in the Future | Digital Breast Tomosynthesis Willingness to be Screened in the Future | Ab-MRI Future Screen if AB-MRI Detects More Cancer Than Mammography or Ultrasound | DBT Future Screen if DBT Detects More Cancer Than Mammography or Ultrasound
Number analyzed (Participants) | 1314 | 1313 | 1319 | 1318
Participants
  Screen every year | 1107 | 1221 | 1237 | 1271
  Screen every two years | 147 | 66 | 64 | 35
  Screen every three years | 34 | 13 | 7 | 3
  Screen every four Years | 13 | 5 | 4 | 4
  Never Again | 13 | 8 | 7 | 5

7. Secondary Outcome: Factors Associated With Willingness to Return for Screening
Description: Polytomous logistic regression will be used to examine factors associated with willingness to return, including screen result, cancer status, and demographic characteristics.
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2024-12

8. Secondary Outcome: Oncotype-DCIS Scores by Modality
Description: Descriptive Analyses presenting the the distributions of Oncotype-DCIS scores by modality: Ductal carcinoma in situ (DCIS) detected on abbreviated breast-magnetic resonance (MR) and digital tomosynthesis mammography (DBT) A low risk score is less than 39, and a high risk score is 55 or higher. A score of 39 to 54 is intermediate risk.
Time Frame: Up to 1 year
Population: All subjects with DCIS detected either by AbMRI or DBT received Oncotype DX assessment
Measure: Count of Participants; unit: Participants
Groups:
- Digital Breast Tomosynthesis (DBT) Oncotype DX for DCIS: Oncotype DX results for Digital Breast Tomosynthesis (DBT) DCIS. Imaging performed within 30 days following registration.
  DBT and abbreviated -MR were performed on the same day and interpreted by two different radiologists, each blinded to the other modality. However, DBT and AB-MR were allowed to be performed within 24 hours of each other, as long as the radiologists remained blinded to the results of the other modality
- Abbreviated Breast MR (AB-MR) Oncotype DX for DCIS: Oncotype DX results for abbreviated breast MR (AB-MR) detected DCIS. Imaging performed within 30 days following registration.
  DBT and AB-MR were performed on the same day and interpreted by two different radiologists, each blinded to the other modality. However, DBT and AB-MR were allowed to be performed within 24 hours of each other, as long as the radiologists remained blinded to the results of the other modality
Arm/Group | Digital Breast Tomosynthesis (DBT) Oncotype DX for DCIS | Abbreviated Breast MR (AB-MR) Oncotype DX for DCIS
Number analyzed (Participants) | 10 | 10
Participants
  Low (<39) | 1 | 2
  Intermediate (39-54) | 0 | 1
  High risk (>54) | 0 | 0
  Tissue not available/not submitted | 4 | 3
  DCIS not detected by Modality | 5 | 4

9. Secondary Outcome: Incident Cancer Rate
Description: Breast cancer incidence will be estimated. Person-years will be measured.
Time Frame: Up to 3 years
Population: All eligible subjects who received both Ab-MR and DBT at year 0 and year 1
Measure: Number (95% Confidence Interval); unit: cancers per 1,000 person-years
Groups:
- All Participants: All participants scheduled for both DBT and AB-MR Estimated incident cancer rate (95% CI): interpreted as number of incident cancers per 1,000 person-years
Arm/Group | All Participants
Number analyzed (Participants) | 1291
cancers per 1,000 person-years
  Year 1 Screen to 12 mo post screening | 7.89 [3.79 to 14.52]
  12 months to 24 months post study screening | 3.19 [0.87 to 8.18]
  24 months to 36 months study screening | 5.00 [1.84 to 10.89]

10. Secondary Outcome: NanoString Tumor Biologies of Invasive Cancers and Ductal Carcinoma in Situ (DCIS) Detected on AB-MR and DBT
Description: For all invasive cancers detected during the study period, the NanoString PAM50 will be performed. The frequencies of cancer types determined by the NanoString analysis will be tabulated and compared. For DCIS, if the Oncotype-DCIS score was performed, the distributions of scores will be tabulated and compared.
  All efforts to obtain NanoString data have been exhausted, therefore we have no data available to report.
Time Frame: end of study
Population: NanoString data were not collected
Groups:
- Digital Breast Tomosynthesis (DBT) PAM50 NanoString for DCIS: PAM50 NanoString results for Digital Breast Tomosynthesis (DBT) DCIS. Imaging performed within 30 days following registration.
  DBT and abbreviated -MR were performed on the same day and interpreted by two different radiologists, each blinded to the other modality. However, DBT and AB-MR were allowed to be performed within 24 hours of each other, as long as the radiologists remained blinded to the results of the other modality
- Abbreviated Breast MR (AB-MR) PAM50 NanoString for DCIS: PAM50 NanoString results for abbreviated breast MR (AB-MR) detected DCIS. Imaging performed within 30 days following registration.
  DBT and AB-MR were performed on the same day and interpreted by two different radiologists, each blinded to the other modality. However, DBT and AB-MR were allowed to be performed within 24 hours of each other, as long as the radiologists remained blinded to the results of the other modality
Arm/Group | Digital Breast Tomosynthesis (DBT) PAM50 NanoString for DCIS | Abbreviated Breast MR (AB-MR) PAM50 NanoString for DCIS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year for Adverse Events and All deaths while on-study
Description: Serious Adverse Events (SAE), in addition to the standard definition include:
  All Grade 5 events occurring within 30 days of imaging, regardless of attribution or unexpectedness All Grade 4 events occurring within 30 days of imaging that are unexpected and have an attribution of "Possible, Probable, Definite" All Grade 4 kidney adverse events All occurrences of Nephrogenic Systemic Fibrosis (NSF) or Nephrogenic Fibrosing Dermopathy (NFD) All Grade 5 events while on study
Groups:
- All Participants: All participants scheduled for both DBT and AB-MR Note, because of the temporal proximity (generally the same day), it is not possible to attribute the adverse events either by arm or by an individual modality.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 6/1444
Serious Adverse Events (participants affected / at risk) | 6/1444
Other Adverse Events (participants affected / at risk) | 25/1444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=1444)
Death NOS (General disorders) | 3 (3) — Death not otherwise specified [NOS] occurring more than 461 days after the year 0 screening intervention.
Disease progression (General disorders) | 1 (1) — Disease progression [Death] This death occurred 395 days after the year 0 screening intervention and after hospital admission for neurosurgery for metastatic disease to the brain.
Malignant neoplasm of the right lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Malignant neoplasm of the right lung [Death] occurring 136 days after the year 0 screening intervention.
Intracranial hemorrhage (Nervous system disorders) | 1 (1) — Intracranial hemorrhage [Death] occurring 106 days after the year 0 screening intervention.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory failure [Death] This death occurred 395 days after the year 0 screening intervention and after hospital admission for neurosurgery for metastatic disease to the brain.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=1444)
Vertigo (Ear and labyrinth disorders) | 1 (1) — Vertigo [Mild symptoms]
Bilateral Eye swelling (Eye disorders) | 1 (1) — Bilateral Eye swelling [Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; no change in vision]
Nausea (Gastrointestinal disorders) | 2 (2) — Nausea [Loss of appetite without alteration in eating habits]
Vomiting (Gastrointestinal disorders) | 1 (1) — Vomiting [3 - 5 episodes (separated by 5 minutes) in 24 hrs]
Facial rash (General disorders) | 1 (1) — Facial rash [Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated]
Infusion site extravasation (General disorders) | 1 (1) — Infusion site extravasation [Painless edema]
Localized edema (General disorders) | 1 (1) — Localized edema [Moderate localized edema and intervention indicated; limiting instrumental ADL]
Pain (General disorders) | 1 (1) — Pain [Mild pain]
Allergic reaction (Immune system disorders) | 2 (2) — Allergic reaction [Intervention or infusion interruption indicated; responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics); prophylactic medications indicated for <=24 hrs]
Allergic reaction (Immune system disorders) | 1 (2) — Allergic reaction [Transient flushing or rash, drug fever <38 degrees C (<100.4 degrees F); intervention not indicated]
Bruising (Injury, poisoning and procedural complications) | 1 (1) — Bruising [Localized or in a dependent area]
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) — Vascular access complication [Device dislodgement, blockage, leak, or malposition; device replacement indicated]
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Back pain [Mild pain]
Vasovagal reaction (Nervous system disorders) | 2 (2) — Vasovagal reaction [Present]
Anxiety (Psychiatric disorders) | 2 (2) — Anxiety [Mild symptoms; intervention not indicated]
Breast pain (Reproductive system and breast disorders) | 1 (1) — Breast pain [Moderate pain; limiting Instrumental activities of daily living (IADL)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Cough [Mild symptoms; nonprescription intervention indicated]
Flushing (Vascular disorders) | 1 (1) — Flushing [Asymptomatic; clinical or diagnostic observations only; intervention not indicated]
Hematoma (Vascular disorders) | 1 (1) — Hematoma [Mild symptoms; intervention not indicated]
Hematoma (Vascular disorders) | 1 (1) — Hematoma [Minimally invasive evacuation or aspiration indicated]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT02933489/Prot_SAP_001.pdf
  • Informed Consent Form (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT02933489/ICF_000.pdf